CLINICAL TRIAL: NCT01932723
Title: Effect of Functional Lumbar Stabilization Exercises on Pain, Disability and Kinesiophobia in Women With Menstrual Low Back Pain
Brief Title: Effect of Functional Lumbar Stabilization Exercises in Women With Menstrual Low Back Pain
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Amir Massoud Arab, Dr., University of Social Welfare and Rehabilitation Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 891025
Record Dates: First submitted 2013-06-26; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain
Keywords: Stabilization exercises, Pain, Disability, Menstruation
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumbar Stabilization Exercises & Control (Experimental): Lumbar stabilization exercises daily, 10 repetitions each (three times a day) for three months consecutively. All exercises were performed to a count of 7 seconds.
  Interventions: Behavioral: Lumbar stabilization exercises

INTERVENTIONS:
Behavioral: Lumbar stabilization exercises — The functional lumbar stabilization exercises was performed daily, 10 repetitions each, three times a day for three months consecutively.
  Other Names: Trunk stabilization exercice, Stability exercise

SUMMARY:
Menstrual low back pain (LBP) is one of the common complaints among women. Menstrual LBP may be attributed to the spinal instability resulting from ligament laxity due to hormonal change. The purpose of this study was to investigate the effect of functional lumbar stabilization exercises on pain, disability and kinesiophobia in women with menstrual LBP.

DETAILED DESCRIPTION:
Pain intensity using Numeric Pain Scale (NPS), Oswestry disability index (ODI), Roland-Morris questionnaire (RMQ) and Tampa scale of kinesiophobia (TSK) were collected at base line and at the end of treatment (after three months) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain LBP during menstrual phase (days 1-6) of the menstrual cycle.
* Suffering from low back pain during all menstrual cycles in the year before the study.
* No back pain or low back paiun at times other than the menstrual phase.
* Pain intensity during menstrual LBP greater than 5 in Numeric Pain Scale

Exclusion Criteria:

* History of spinal surgery, spinal or pelvic fracture and hospitalization for severe trauma or car accident, urinary tract infection, vaginal infection and known neurological disorders.
* Pain intensity lesser than 5 in Numeric Pain Scale

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pain | one year
  Pain intensity using Numeric Pain Scale (NPS) were collected at base line and at the end of treatment.

SECONDARY OUTCOMES:
Disability | One year
  Oswestry disability index (ODI) and Roland-Morris questionnaire (RMQ) were collected at base line and at the end of treatment.

OTHER OUTCOMES:
Kinesiophobia | One year
  Tampa scale of kinesiophobia (TSK) were collected at base line and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Arab, PhD, Principal Investigator — University of Social Welfare and Rehabilitation Sciences
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Tehran Province, Iran